CLINICAL TRIAL: NCT04542772
Title: Effectiveness of Patient Education on Mirror Therapy to Improve Upper Extremity Function in Acute Stroke Patients
Brief Title: Mirror Therapy Education for Acute Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Health Sciences North Research Institute (Other)
Collaborators: NORTHERN ONTARIO ACADEMIC MEDICINE ASSOCIATION (NOAMA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: C-20-15
Record Dates: First submitted 2020-08-26; First posted 2020-09-09 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy + Standard of Care (Experimental): Participants in this group will receive standard of care based on their needs along with mirror therapy education.
  Interventions: Other: Mirror Therapy; Other: Regular Rehabilitation
- Standard of Care (Active Comparator): Participants in this group will receive only standard of care based on their needs.
  Interventions: Other: Regular Rehabilitation

INTERVENTIONS:
Other: Mirror Therapy — Participants will receive the standard-of-care; multidisciplinary rehabilitation intervention based on their needs and tolerance, and will receive an additional 30 min of Mirror Therapy education. During Mirror Therapy education, the patients will be educated or shown how to perform MT and the patients will complete the recommended exercises on their own for 30 minutes/day for 5 days a week/ for 4 weeks. Standard Mirror Therapy Protocol will be followed.
  Arms: Mirror Therapy + Standard of Care
Other: Regular Rehabilitation — Participants will receive the standard-of-care, multidisciplinary rehabilitation intervention based on their needs and tolerance.

SUMMARY:
In Canada, the number of stroke survivors is equivalent to the size of one of the four Atlantic Provinces. The incident rate of stroke has been increasing steadily since 1995. The majority of the stroke survivors lose upper extremity function, resulting in diminished activities of daily living (ADL). Many therapeutic interventions are recommended to improve upper extremity function or ADLs of stroke survivors, however, Mirror Therapy (MT), inexpensive intervention, can be self-administered by stroke survivors with intact cognition. Thus, the research question is whether a self-administered MT technique improves acute stroke patients' upper extremity motor function and recovery?

ELIGIBILITY:
Inclusion Criteria:

* Admitted with diagnosis of stroke with onset within two weeks
* Medically stable
* Able to follow directions
* No severe cognitive impairments that could interfere with patient participation
* Consent to treatment by patient
* Alpha-Functional Independence Measure (Alpha-FIM) score of > 40

Exclusion Criteria:

* Medical instability
* Lack of motivation
* Recurrent/ chronic stroke
* Recent upper extremity musculoskeletal injuries with movement restrictions
* Receptive or global aphasia
* Delirium
* Unilateral neglect
* Visual field deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment scale | Assessment will be completed at 2 points: Pre-test assessment will be done within 48 hours of stroke admission and post-test assessment will be done at 4 weeks.
  Scores of < 31 corresponded with 'no to poor' upper extremity capacity, 32 to 47 represented 'limited capacity', 48 to 52 represented 'notable capacity' and 53 to 66 represented 'full' upper extremity capacity.
Wolf Motor Function Test | : Assessment will be completed at 2 points: Pre-test assessment will be done within 48 hours of stroke admission and post-test assessment will be done at 4 weeks
  Assess upper extremity function; maximum Score is 75; lower scores are indicative of lower functional levels.

SECONDARY OUTCOMES:
Modified Barthel Index | : Assessment will be completed at 2 points: Pre-test assessment will be done within 48 hours of stroke admission and post-test assessment will be done at 4 weeks
  Assess Activity of Daily Living, Scores of <15 usually represents moderate disability and <10 usually represents severe disability.

REFERENCES:
- [Derived] Rajendran V, Jeevanantham D, Lariviere C, Singh RJ, Zeman L, Papuri P. Effectiveness of self-administered mirror therapy on upper extremity impairments and function of acute stroke patients: study protocol. Trials. 2021 Jul 9;22(1):439. doi: 10.1186/s13063-021-05380-9. PMID 34243808